CLINICAL TRIAL: NCT04684628
Title: Investigation of the Sensitivity and Specificity of 68Ga-HBED-CC-PSMA PET/CT in Prostate Cancer
Brief Title: 68Ga-PSMA PET/CT in Prostate Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is suspended due to some logistic issues
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Rajan Rakheja, Assistant Professor, University of Saskatchewan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PSMA-01
Record Dates: First submitted 2020-12-14; First posted 2020-12-24 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: There will be two groups depending upon the disease status. Cohort 1- Participant will be in Cohort 1 if have biochemical reoccurrence (post-prostatectomy or post radical radiotherapy) or have biochemical relapse with rising PSA in spite of taking hormone treatment (this situation is characterized as non-metastatic castration resistant prostate cancer M0CRPC).
  Cohort 2- Participant will be in Cohort 2 if have high risk prostate cancer and have not received any definitive treatment.
  Participants of both cohorts will receive the same study drug for imaging procedure. Participants of both the cohort will undergo one PET/CT scan at 45 minute after a single dose injection of 68Ga-PSMA-11.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biochemical Reoccurrence (Experimental): Patients with biochemical reoccurrence (post-prostatectomy or post radical radiotherapy) or patients with biochemical relapse with rising PSA in spite of taking hormone treatment (this situation is characterized as non-metastatic castration resistant prostate cancer M0CRPC) and compare it to bone scan and CT in 2 groups:
  PSA >= 0.2 ng/mL and <= 0.5 ng/mL or PSA > 0.5 ng/ml
  Interventions: Drug: 68Ga-PSMA PET/CT
- High Risk Prostate Cancer (Experimental): Patients with high risk prostate cancer who have not received any definitive treatment. These high-risk patients are defined using the D'Amico Classification System: Those with a PSA of more than 20, or a Gleason score equal to or greater than 8, or have a clinical stage greater than T2c.
  Interventions: Drug: 68Ga-PSMA PET/CT

INTERVENTIONS:
Drug: 68Ga-PSMA PET/CT — Administration of 68Ga-PSMA-11 followed by a PET/CT scan at 45 min after injection.

SUMMARY:
This is a single-center, multi-arm, open-label, phase III trial in up to 500 patients with biopsy-proven prostate cancer.

Participants will receive regular standard of clinical care. The only study-specific procedures will the administration of 68Ga-PSMA-11 followed by a PET/CT (positron emission tomography/computed tomography) scan. Participants will be followed for two hours after the infusion for identification of any immediate adverse events (AE), and will be contacted by telephone after 7 to 14 days to enquire about any delayed AEs.

PET/CT images, CT-alone images and bone scans will be read by separate readers who will not be blinded to all other clinical and imaging information. The standard of truth will be a consensus of the readers based on all available clinical, imaging, and histopathological information available for up to 6 months after the PET/CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18 years or older
* Previously diagnosed with prostate cancer, under referring physician's care
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine (or prone) for up to 40 minutes and tolerating intravenous cannulation for injection

Exclusion Criteria:

* Patients who are medically unstable (e.g. acute cardiac or respiratory distress or hypotensive)
* Patients who exceed the safe weight limit of the PET/CT bed (usually approximately 400 lbs.) or who cannot fit through the PET/CT bore (usually approximately 70 cm diameter)
* Patients with unmanageable claustrophobia

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male participant previously diagnosed with prostate cancer, under referring physician's care.
Enrollment: 500 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 68Ga-PSMA-11 PET/CT compared to that of CT alone and bone scan in two different cohorts of prostrate cancer patients. | 6 months
  PET/CT images, CT-alone images and bone scans will be read by separate readers who will not be blinded to all other clinical and imaging information. A target lesion list will be created, finalized and entered into the research study file. Reviewer will assign each patient an overall likelihood of prostate cancer score, equal to the highest score of any target lesion on the PET/CT scan. Following the entry of final PET/CT, CT-only and bone scan target lesion lists and overall likelihood scores into the study file, all the experienced readers will become un-blinded and adjudicate by consensus in conjunction with referring physicians all lesions identified by each on their respective datasets and will assign a final consensus to each lesion. Each target lesion identified by each reader will be followed clinically, radiologically and histopathologically over a minimum period of 6 months and the final consensus can be modified based on this follow-up.

SECONDARY OUTCOMES:
The secondary endpoint is the number of adverse events, both immediate and delayed. | baseline (i.e. Imaging visit) and at the end of study visit (day 7 to day 14)
  Immediate and delayed adverse events will be captured for every patient and will be analysed at the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Rakheja, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada